CLINICAL TRIAL: NCT06207279
Title: Preliminary Study on the Development and Reliability and Validity of Attention Rating Scale
Status: Recruiting | Type: Observational
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Xueqin Wang, Principle Investigator, Peking University Sixth Hospital
Other Study IDs: 2022-056
Record Dates: First submitted 2023-10-10; First posted 2024-01-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Depression; Insomnia; Attention Disturbances; Healthy
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Major Depressive Disorder: Patients meeting the diagnostic criteria for Major Depressive Disorder (MDD) according to DSM-5.
  Interventions: Diagnostic Test: rating
- Chronic Insomnia Disorder: Patients meeting the diagnostic criteria for Chronic Insomnia Disorder according to ICSD-3.
  Interventions: Diagnostic Test: rating
- Health Control: Healthy population.
  Interventions: Diagnostic Test: rating
- Attention Deficit and hyperactivity Disorder: Patients meeting the diagnostic criteria for Attention Deficit and hyperactivity Disorder (ADHD) according to DSM-5.
  Interventions: Diagnostic Test: rating

INTERVENTIONS:
Diagnostic Test: rating — rating scales, test ANT

SUMMARY:
This study, based on preliminary experimental results, literature review, and expert consultations, developed the Attentional Rating Scale (ARS). The aim was to rapidly assess participants' attention and potential influencing factors. The research focused on the scale's reliability and validity among healthy adults. Additionally, the Attention Network Test (ANT) served as the gold standard for evaluating attention. The study attempted to identify correlations between various dimensions of attention and the three attentional networks.

DETAILED DESCRIPTION:
1. To adiministrate 60 healthy subjects to evaluate internal consistency reliability.
2. To choose 20 cases for ARS retesting 7 days after the first ARS evaluation.
3. To evaluate the split half reliability through the Spearman Brown coefficient.
4. To apply principal component analysis for structural validity analysis.
5. Using the Attention Network Test (ANT) and Toronto Hospital Alertness Test (THE) as gold standards, the Pearson correlation coefficient was used for criterion validity analysis.
6. To administrate 60 patients with MDD, ADHD and insomnia disorder testing the discrimination validity of ARS.

ELIGIBILITY:
Inclusion Criteria:

1. Major Depressive Disorder (MDD) or attention deficit hyperactivity disorder (ADHD) diagnosed according to DSM-5, or Chronic Insomnia Disorder diagnosed according to ICSD-3
2. Ages between 18 and 60 years old
3. Right-handed
4. Educational level ≥5 years or IQ ≥90, capable of understanding and reading Chinese.

Exclusion Criteria:

1. Currently diagnosed with any other DSM-5 mental disorders (according to MINI 7.0) or ICSD-3 sleep-wake disorders, apart from MDD, ADHD or insomnia disorder
2. Currently and past history of neurological disorders and physical illnesses with subjectives
3. Consumed alcohol in the week preceding the enrollment
4. Using antidepressants, antipsychotics, mood stabilizers, or other central nervous system-acting drugs for at least 4 weeks in the current episode
5. Undergoing any physical treatments such as ECT, neuromodulation therapy or Traditional Chinese Medicine treatment in the past 6 months
6. Refused to sign the informed consent form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixty cases of patients diagnosed with Major Depressive Disorder (MDD), ADHD and insomnia disorder separately are recruited from outpatient clinics and hospital wards. Additionally, sixty healthy individuals are recruited from the community as control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Developing Attention Rating Scale（ARS） | 3 months
  The Attention Assessment Scale is developing as a tool to assess attention ability designed for self-rating scale. Its purpose is to swiftly evaluate the attention levels of adults. There are 30 items in ARS. The minimum value is 1 and maximum value is 5, and the higher scores mean a better outcome for attention ability.
Reliability and Validity of the Attention Assessment Scale. | 2 years
  Reliability
  1. Cronbach α of ARS should be above 0.8 that means good reliability.
  2. The intra group correlation value for retesting reliability should be above 0.8 that means good retesting reliability.
  Validity
  1. The split half reliability measured and factor analysis to test constuctive validity of ARS.
  2. The correlation coefficient r with ANT and the correlation coefficient r with THAT should be statistic significant, that means good validity of attention ability for Attention Assessment Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqin Wang, doctor, Principal Investigator — Peking University Sixth Hospital
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No